CLINICAL TRIAL: NCT06597279
Title: Developing Tools for Dialysis Decision Support
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Palo Alto Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Manjula Kurella Tamura, MD, MPH, Nephrologist and clinical investigator, VA Palo Alto Health Care System
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB-54542; HX002763 (Other Grant/Funding Number: VA HSRD)
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: This is a non-randomized controlled trial using historical control as a comparator. It involves comparing outcomes from a group of participants receiving the current intervention with outcomes from a previously treated group (historical control) that did not receive the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Web-based dialysis decision support tool
  Interventions: Behavioral: Web-based dialysis decision support tool
- Control (No Intervention): Historical controls

INTERVENTIONS:
Behavioral: Web-based dialysis decision support tool — The intervention in this study is the "Kidney Care Roadmap", a web-based dialysis decision support tool designed to assist patients with advanced chronic kidney disease and their caregivers.
  Arms: Intervention

SUMMARY:
The aim of this study is to evaluate the impact of a web-based dialysis decision support tool on decisional conflict, and values-treatment concordance and other decisional outcomes in individuals with advanced chronic kidney disease, and to assess the tool's acceptability and usability.

DETAILED DESCRIPTION:
This study employs a pre-post design to assess the impact of a web-based dialysis decision support tool on patients with advanced chronic kidney disease and their caregivers. Participants will complete baseline surveys assessing demographics, knowledge of kidney failure treatments, and decisional conflict during a nephrology clinic visit. Following the visit, participants will access the decision support tool, with follow-up support provided by the study coordinator. One to four weeks after the baseline visit, participants will complete follow-up surveys to re-evaluate knowledge, decisional conflict, values-treatment concordance, and the quality of shared decision-making. Additionally, telephone interviews will be conducted to explore participants' understanding of treatment options and gather feedback on the decision support tool.

ELIGIBILITY:
Inclusion Criteria:

1. Age >=65
2. Estimated GFR <25 ml/min/1.73m2
3. English speaking
4. Not a candidate for kidney transplant based on nephrologist assessment.

Family/caregiver inclusion criteria:

1. age >=21
2. English speaking

Exclusion Criteria:

a. Patients with cognitive impairment will be excluded; however their family member or caregiver is eligible to participate.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-11-21 (Actual); Primary Completion 2025-04-10 (Actual); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Treatment choice | 1 month
  Proportion of patients who are undecided about treatment choice.
Values treatment concordance | 1 month
  Change in values treatment concordance.
Confidence in treatment decision | 1 month
  Confidence in kidney failure treatment decision
Treatment choice | 1 month
  Proportion of patients who choose medical management without dialysis
Decisional Conflict Scale (DCS) | 1 month
  Change in the decisional conflict scale (DCS) score from baseline to follow-up. Scores range from 0 [no decisional conflict] to 100 [extremely high decisional conflict].

CONTACTS AND LOCATIONS:
Overall Officials: Manjula Tamura, MD, MPH, Principal Investigator — U.S. Department of Veterans Affairs - Palo Alto Health Care System
Locations (2):
- United States (2):
  - U.S. Department of Veterans Affairs - Palo Alto Health Care System, Palo Alto, California
  - Stanford Health Care, Stanford, California

IPD SHARING:
Plan to Share IPD: No